CLINICAL TRIAL: NCT00521807
Title: Hypnosis as a Treatment of Chronic Widespread Pain in General Practice. A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26035831907
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2007-08

CONDITIONS: Chronic Widespread Pain
Keywords: Hypnosis,; Chronic widespread pain,; CWP,; General Practice
MeSH Terms: conditions — Chronic Pain | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 1 (No Intervention)
- A 2 (Experimental): Treatment group
  Interventions: Procedure: Hypnosis

INTERVENTIONS:
Procedure: Hypnosis — a standardized hypnosis treatment with ten consecutive therapeutic sessions once a week,
  Arms: A 2

SUMMARY:
Objective: The study was performed to evaluate the effect of a standardized hypnosis treatment used in general practice for patients with chronic widespread pain (CWP).

Design: A randomized control group-controlled study. Setting and subjects: 16 patients were randomized into a treatment group or a control group, each constituting eight patients. Seven patients in the treatment group completed the schedule. After the control period, five of the patients in the control group also received treatment, making a total of 12 patients having completed the treatment sessions.

Intervention: The intervention group went through a standardized hypnosis treatment with ten consecutive therapeutic sessions once a week, each lasting for about 30 minutes, focusing on ego-strengthening, relaxation, releasing muscular tension and increasing self-efficacy.

Main outcome measures: A questionnaire was developed in order to calibrate the symptoms before and after the 10 weeks period, and the results were interpolated into a scale from 0 to 100, increasing numbers representing increasing suffering.

ELIGIBILITY:
Inclusion Criteria:

* Chronic widespread pain for at least three months and at most five years.

Exclusion Criteria:

* Patients having primarily other organic diseases or serious psychiatric disorders were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2001-03; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan R Grondahl, Dr, Principal Investigator — The Institute of General Practice and Community Medicine, University of Oslo, Norway.
Locations (1):
- 1) Institute of General Practice and Community Medicine, University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Grondahl JR, Rosvold EO. Hypnosis as a treatment of chronic widespread pain in general practice: a randomized controlled pilot trial. BMC Musculoskelet Disord. 2008 Sep 18;9:124. doi: 10.1186/1471-2474-9-124. PMID 18801190